CLINICAL TRIAL: NCT02317250
Title: Early and Long-Term Health Outcomes of Molecular Cerebral Imaging in Incipient Dementia (MCI-ID) II
Brief Title: Molecular Cerebral Imaging in Incipient Dementia (MCI-ID) II
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study withdrawn. No participants enrolled.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel H. Silverman, Professor, Medical and Molecular Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 11-00815-02
Record Dates: First submitted 2014-12-09; First posted 2014-12-15 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's disease; Alzheimer disease; MDC; Mild Decline in Cognition; MCI; Dementia; PET; FDG-PET; FDG; amyloid; amyloid imaging; CMS; Coverage with Evidence Development; CED; MCI-ID
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- prompt amyloid imaging, delayed FDG-PET (Experimental): Subject's managing physicians will be given the results of amyloid imaging scans immediately. FDG-PET results will be released two years after scanning.
  Interventions: Procedure: Amyloid imaging; Procedure: FDG-PET
- prompt FDG-PET, delayed amyloid imaging (Experimental): Subject's managing physicians will be given the results of FDG-PET scans immediately. Amyloid imaging results will be released two years after scanning.
  Interventions: Procedure: Amyloid imaging; Procedure: FDG-PET
- prompt FDG-PET, prompt amyloid imaging (Experimental): Both FDG-PET and amyloid imaging scan results will be made immediately available to the managing physician.
  Interventions: Procedure: Amyloid imaging; Procedure: FDG-PET
- delayed FDG-PET, delayed amyloid imaging (Active Comparator): Neither FDG-PET nor amyloid imaging scan results will be released to the managing physician for 2 years.
  Interventions: Procedure: Amyloid imaging; Procedure: FDG-PET

INTERVENTIONS:
Procedure: Amyloid imaging — Amyloid imaging brain scans are administered once to all arms.
Procedure: FDG-PET — [F-18] FDG-PET brain scans are administered once to all arms.

SUMMARY:
A substantial portion of people covered by Medicare will develop Alzheimer's disease and other forms of dementia that together devastate the lives of millions of people in the United States, and cost us a total of over $200 billion every year. Getting a brain scan with a PET scanner to look for abnormal brain metabolism patterns is recognized as "reasonable and necessary" for some patients with "a recently established diagnosis of dementia" (Centers for Medicare and Medicaid Services (CMS), Decision Memo CAG-00088R), but the evidence is considered less clear for patients having less severe cognitive problems, and/or for patients getting a brain scan with a PET scanner to look for abnormal proteins in the brain (CMS Decision Memo CAG-00431N). This project employs a scientifically rigorous design (prospective, multi-centered, randomized controlled trial) to determine whether such PET scanning can help distinguish more accurately than is being done in current clinical practice those patients with early molecular changes in their brains who will benefit from Alzheimer related treatments from those patients who will not, as proven by measuring to what extent the PET scans actually lead to earlier appropriate therapy, and in fact result in improved outcomes for Medicare beneficiaries and for the health care system in which they obtain care.

DETAILED DESCRIPTION:
The overarching objective of this project is to test whether diagnostic assessments informed by data on molecular cerebral changes can lead to improved health outcomes of an epidemiologically major segment of the geriatric patient population - people experiencing changes in their cognitive skills relative to their prior level of cerebral functioning. In the present proposal, we specifically aim to measure how knowledge of molecular cerebral information 1) influences the therapeutic management of patients being evaluated for symptoms of cognitive decline, and 2) impacts upon long-term health outcomes, particularly for patients having findings on positron emission tomography (PET) scans consistent with presence of Alzheimer's disease (AD)- like changes in their brains. Patients suffering from documentable decline of cognitive function will undergo baseline neuropsychologic testing, and neuroimaging with MRI and PET. Reports of PET scans will be sealed at the time of interpretation, and then randomized with respect to whether they are released to the patients' managing physicians at the time of interpretation, or two years after the time that scanning is performed. All treatment decisions will be made by the managing physicians and their patients. Cognitive abilities, functional status, and other clinical and social history parameters will be assessed every six months. Our central hypothesis is that among the group of patients whose PET scan results are conveyed to their physicians at the time of scanning, cognitive and functional abilities will be maintained at a higher level during the two years following PET. Beyond addressing the specific aims noted above and further described below, a valuable feature of this project will be the collection of a rich source of data that can be used to address many questions beyond its major focus (e.g., diagnostic value of volumetric MRI data used instead of, or in conjunction with, PET data in the Medicare beneficiary population; incremental value of applying statistically parameterizing and/or quantifying software tools to PET data). The protocol has been designed to conform to all standards specified by the Centers for Medicare and Medicaid Services (CMS) for Coverage with Evidence Development (CED), generally, and with all requirements for a CED study responsive to CMS Decision Memo CAG-00431N, specifically.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive decline and/or personality change is present, as observable by physician and/or close contact(s) of the patient; or in the absence of this, the patient provides a clear history of decline that the patient's physician deems to be reliable.
2. If history or neurologic exam reveals findings suspicious for stroke, tumor, bleed, ictal activity, or hydrocephalus, then CT/MRI and appropriate neurological or neurosurgical consultation must have been obtained.
3. Standard history, physical, and laboratory screen have been performed to identify possible presence of depression, substance abuse, malnourishment, medication effects and interactions, cardiopulmonary compromise, electrolyte/calcium imbalance, anemia, hypoxemia, infection, thyroid dysfunction, renal dysfunction, hepatic dysfunction, or glucose dysregulation.
4. Any positive findings revealed in 2) or 3) above have been appropriately treated, wherever possible, but cognitive/behavioral deficit persists post-therapy.

Exclusion Criteria:

1. Subjects under age 65 will not be recruited, in order to enhance the relevance of the project by focusing on the group of Medicare beneficiaries in whom serious concerns about early signs and symptoms of senile onset dementia are most typically emerging.
2. Cognitive dysfunction has impaired subject's ability to perform activities of daily living.
3. Present or past history of thyroid disease.
4. Claustrophobia or metal in body or other condition that would preclude PET or MRI from being acquired.
5. Visual, auditory or motor deficits that would preclude accurate neuropsychological testing.
6. AD-specific pharmacotherapy already initiated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Rate of change from baseline in neuropsychological (cognitive,functional) test results | baseline, 6 months, 12 months, 18 months, 24 months
  Study participants will undergo neuropsychological testing at baseline and every six months for two years.
Utilization of healthcare resources | over 2 years
FDG-PET and amyloid imaging results, compared with working diagnoses made before and after time of imaging | baseline and up to 2 years
  Study participants will undergo FDG-PET and amyloid imaging. Working diagnoses made before and after the imaging is performed will be compared.
Rates of prescription of AD-specific therapies | baseline, 6 months, 12 months, 18 months, 24 months
  Comparisons between the rate of prescription for AD-specific therapies and release type (either immediate or delayed release) will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Silverman, MD, Ph.D., Principal Investigator — University of California, Los Angeles